CLINICAL TRIAL: NCT02777502
Title: Effects of Cannabidiol on Marijuana-seeking in Humans
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Other Study IDs: CBD-1
Record Dates: First submitted 2016-02-11; First posted 2016-05-19 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the proposed study is to investigate the effectiveness of cannabidiol for reducing marijuana seeking in non-treatment seeking volunteers. Cannabidiol is a cannabinoid (similar to cannabis, or marijuana) present in marijuana that alters some of the effects of marijuana.

Assess the ability of acute smoked CBD pretreatment to reduce marijuana-seeking behavior and increase price-elasticity of marijuana demand.

DETAILED DESCRIPTION:
Participants will be asked to participate in a total of three choice sessions over two weeks with each session day separated by at least two days. Each session day will last approximately 8 hours.

During each study session participants will be asked to smoke a cigarette. Participants will be asked to smoke from a marijuana cigarette. These cigarettes may contain cannabidiol or they may not (placebo).

Participants will be asked to answer questions about how the drugs make them feel. Vitals signs (blood pressure, heart rate, and oxygen saturation) will be measured using a non-invasive (external) vitals monitor.

Six samples will be taken in each of the three sessions. Blood samples will be obtained via butterfly catheter placed in a vein.

Participants will be asked to remain in the laboratory until all marijuana-related subjective and physiological effects have returned to the original levels recorded this morning before they smoked the first marijuana cigarette.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be males and females aged 21-45 yrs.
2. Must be in generally good health.
3. Volunteers may meet DSM-5 criteria for current Cannabis Use Disorder but not currently be in treatment or seeking treatment for their substance use problems.
4. An observed, temperature-tested urine specimen must test positive for THC so that inclusion is not solely based on self-report.

Exclusion Criteria:

1. Psychiatric illness other than Cannabis or Nicotine Use Disorder. Also exclusionary is a history or suspicion of psychosis or indication of behavior not conducive to compliance with the study protocol.
2. Neurologic disease: structural brain abnormalities (e.g., neoplasms), cerebrovascular disease, seizures, infectious disease, history of other neurological diseases, or head trauma resulting in unconsciousness.
3. Cardiovascular disease: edema, chest pain or palpitations on exertion or drug use, myocardial infarction, systolic blood pressure greater than 160 or less than 95 mmHg, or diastolic pressure greater than 95 mmHg.
4. Pulmonary disease: obstructive pulmonary disease, apnea, cor pulmonale, tuberculosis, dyspnea, orthopnea, or tachypnea (> 24 breaths per minute). Current diagnosis of or treatment for asthma. History of asthma may be allowed, per the study physician's discretion.
5. Systemic disease: e.g., endocrinopathies, renal or hepatic failure, active hepatitis (liver function tests > 3x normal cutoff), myxedema, hypothyroidism, adrenocortical insufficiency, Cushing syndrome, chronic GI disease, AIDS or any other autoimmune disease involving the CNS.
6. Current substance use disorders other than Cannabis or Nicotine Use Disorder.
7. Cognitively impairment as indicated by an estimated IQ of lower than 85. Individuals unable to give voluntary informed consent will not be enrolled. They can be neither intoxicated nor undergoing withdrawal at the time of screening and consent.
8. Recent experimental participation (within past month).
9. Pregnancy or lactation. Females who are heterosexually active and not using (self-report) medically approved birth control measures (e.g., sterilization, tubal ligation, birth control pills, abstinence, intrauterine device, barrier method, cervical cap combined with a spermicide) are not eligible. Women who are breastfeeding will be excluded.
10. Individuals currently in, intending to seek, or court mandated for substance abuse treatment will be excluded. Finally, participants may be withdrawn from study if they do not comply with the study protocol, test positive for drugs of abuse other than marijuana on the routine urine screen or decide not to participate in the study.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Marijuana Dependent Participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Marijuana Craving Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Marijuana Craving VAS administered at baseline 0900. Administered at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 administered every 15 minutes until 1430, then every 30 minutes until 1630.
Marijuana Craving Questionnaire (Self-report measure) | Change is being assessed. Marijuana Craving Quest. administered at baseline 0900. Administered at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 administered every 15 minutes until 1430, then every 30 minutes until 1630.
Marijuana Rating Form (Self-report measure) | Change is being assessed. Marijuana Rating Form administered at baseline 0900. Administered at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 administered every 15 minutes until 1430, then every 30 minutes until 1630.
Subjective Effects Scale Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Subjective Effects Scale administered at baseline 0900. Administered at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 administered every 15 minutes until 1430, then every 30 minutes until 1630.
State-Trait Anxiety Inventory (Self-report measure) | Change is being assessed. State-Trait Anxiety administered at baseline 0900. Administered at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 administered every 15 minutes until 1430, then every 30 minutes until 1630.
Systolic blood pressure (physiological effects) | Change is being assessed. Systolic blood pressure measured at baseline 0900. Then measured at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 measured every 15 minutes until 1430, then every 30 minutes until 1630.
  Examine whether acute smoked cannabidiol (CBD) attenuates physiological (cardiovascular) effects of marijuana.
Diastolic blood pressure (physiological effects) | Change is being assessed. Diastolic blood pressure measured at baseline 0900. Then measured at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 measured every 15 minutes until 1430, then every 30 minutes until 1630.
  Examine whether acute smoked cannabidiol (CBD) attenuates physiological (cardiovascular) effects of marijuana.
Heart rate (physiological effects) | Change is being assessed. Heart rate measured at baseline 0900. Then measured at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 measured every 15 minutes until 1430, then every 30 minutes until 1630.
  Examine whether acute smoked cannabidiol (CBD) attenuates physiological (cardiovascular) effects of marijuana.
Core-body temperature (physiological effects) | Change is being assessed. Core-body temperature measured at baseline 0900. Then measured at 0945 and every 15 minutes until 1045, then every 30 minutes until 1245. At 1330 measured every 15 minutes until 1430, then every 30 minutes until 1630.
  Examine whether acute smoked cannabidiol (CBD) attenuates physiological (cardiovascular) effects of marijuana.
Derive peak concentration (Cmax) | Change is being assessed.Six samples will be taken in each session: prior to the Cannabidiol dose (-15 min), and at 0.5, 1, 2, 3, and 4 h post-Cannabidiol
  Cannabidiol Pharmacokinetics
Time to peak (Tmax) and 6-hr area under the curve (AUC) measures | Change is being assessed.Six samples will be taken in each session: prior to the Cannabidiol dose (-15 min), and at 0.5, 1, 2, 3, and 4 h post-Cannabidiol
  Cannabidiol Pharmacokinetics
Safety of Cannabidiol (CBD) for reducing marijuana seeking in non-treatment seeking volunteers with Cannabis use Disorders | Change is being assessed throughout three 30-minute computer procedures that will be conducted during each of the three choice sessions. The three choice sessions will be conducted over two weeks, with each session day separated by at least 2 days.
  Measure drug-seeking behavior using a computerized (laptop) choice, progressive ratio procedure which allows participant to choose between marijuana puffs or money.
Efficacy of Cannabidiol (CBD) for reducing marijuana seeking in non-treatment seeking volunteers with Cannabis use Disorders | Change is being assessed throughout three 30-minute computer procedures that will be conducted during each of the three choice sessions. The three choice sessions will be conducted over two weeks, with each session day separated by at least 2 days.
  Measure drug-seeking behavior using a computerized (laptop) choice, progressive ratio procedure which allows participants to choose between marijuana puffs or money.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No